CLINICAL TRIAL: NCT05860543
Title: Multi-Institutional Evaluation of C2i-Test Performance for Detecting Molecular Residual Disease (MRD) in Muscle-invasive Bladder Cancer Patients Undergoing Radical Cystectomy.
Brief Title: Clinical Performance Evaluation of the C2i Test
Status: Withdrawn | Type: Observational
Why Stopped: C2i genomics was acquired by veracyte
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, yair lotan, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU-2023-0182
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Muscle Invasive Bladder Cancer
Keywords: C2i-Test; C2i-WGS-MRD Test; Muscle-invasive bladder cancer; MIBC; Whole-genome sequencing; WGS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: C2i-WGS-MRD Test — The C2i-WGS-MRD Test (hereinafter referred to as C2i-Test), a personalized molecular circulating tumor DNA (ctDNA) test, is an in vitro qualitative test that uses next generation sequencing (NGS) based whole-genome sequencing (WGS) data for detecting molecular residual disease (MRD) in patients diagnosed with muscle-invasive bladder cancer (MIBC) and histopathologically classified as stage II-IIIA

SUMMARY:
The overall objective of this study is to demonstrate the safety and effectiveness by means of investigation of the ability of C2i-Test to predict 2-year recurrence-free survival post-RC in stage II-IIIA MIBC patients.

DETAILED DESCRIPTION:
This is a prospective non-interventional study to evaluate the specificity of the C2i-Test in predicting 2-year recurrence-free survival post- definitive treatment (RC/RC + adjuvant chemotherapy), compared to the gold standard (GS) diagnosis as determined by patient outcome (based on NCCN guidelines).

The C2i-WGS-MRD Test (hereinafter referred to as C2i-Test), a personalized molecular circulating tumor DNA (ctDNA) test, is an in vitro qualitative test that uses next generation sequencing (NGS) based whole-genome sequencing (WGS) data for detecting molecular residual disease (MRD) in patients diagnosed with muscle-invasive bladder cancer (MIBC) and histopathologically classified as stage II-IIIA. The C2i-Test is a single site assay performed in the C2i Genomics' CLIA-certified laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have clinically and pathologically confirmed diagnosis of MIBC. Participants with MIBC, path T2-T4a N0/1 at cystectomy with imaging studies confirming no distant disease using cross-sectional imaging of abdomen and pelvis and chest imaging (chest X-ray or computed tomography).
* Variant urothelial histology (e.g., micropapillary, plasmacytoid, sarcomatoid, nested variant, lymphoepithelioid, nested variant) is acceptable. Mixed histology (adenocarcinoma, squamous cell) is acceptable if there is a predominant (>50%) urothelial component.
* Histopathologically confirmed urothelial carcinoma as diagnosed by cystectomy.
* A representative FFPE biopsy specimen (from the -cystectomy specimen) with at least 1 H&E slide and 9 unstained slides, with an associated pathology report must be available.
* Subjects must agree to 8mL blood collection during all visits.
* Treatment plans must include RC. Participant is willing and able to comply with the protocol, including RC, pelvic lymph node dissection (PLND), and prostatectomy (if applicable).
* The patient must be deemed appropriate for RC, PLND, and prostatectomy (if applicable) by his/her oncologist and/or urologist.
* Patient's treatment plan may or may not include neoadjuvant treatment, and/or adjuvant treatment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
* English or Spanish speakers
* Age of Subjects: subjects must be at least 22 years of age and older, or age of majority in their local jurisdiction. There is no upper age limit.
* Ability to understand and the willingness to provide an informed consent

Exclusion Criteria:

* Extravesical urothelial carcinoma (UC) that invades the pelvic and/or abdominal wall for bladder cancer (T4b) as evidenced by imaging.
* Evidence of UC in the urinary tract (ureters, renal pelvis, and urethra) as evidenced by work-up in accordance with NCCN guidelines (e.g., abdominal/pelvic imaging) that includes imaging of upper urinary tract collecting system).
* Patients with mixed histology and <50% urothelial component as evidenced by TURBT pathology.
* Tumors that contain any neuroendocrine/small cell component as evidenced by TURBT pathology.
* Diagnosis of 3 or more synchronous cancers.
* Malignancies other than urothelial cancer within 5 years prior to study entry except those with negligible risk of metastases or death and treated with the expectation of curative outcome (such as: carcinoma in situ of the cervix, basal or squamous cell skin cancer, ductal carcinoma in situ treated surgically with curative intent, papillary thyroid carcinoma, localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse, or incidental prostate cancer [Gleason score ≤ 3 + 4 and PSA < 10 ng/mL] undergoing active surveillance and treatment naïve).
* Per physician discretion: patients with severe or uncontrolled concomitant medical, surgical, or psychiatric disease that could affect compliance with the protocol, the results of the study, or interpretation of the results.
* Individuals who cannot provide consent for their own participation will not be included.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically and pathologically confirmed diagnosis of muscle-invasive bladder cancer stage II-IIIIA will be recruited for the study
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Specificity of the C2i-Test in predicting two-year recurrence-free survival | At 2 years
  Specificity will be derived from a two-by-two summary table of observed counts of positive or negative results by C2i-Test and the relevant GS and defined as: C2i-Test Specificity = True Negative /(True Negative +False Positive )

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lotan, MD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No